CLINICAL TRIAL: NCT02567708
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Crossover Study to Investigate the Efficacy, Safety, and Tolerability of Repeat Doses of Inhaled GSK2269557 in Adults With Persistent, Uncontrolled Asthma
Brief Title: A Study to Investigate the Efficacy, Safety, and Tolerability of Repeat Doses of Inhaled GSK2269557 in Adults With Persistent, Uncontrolled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201543
Record Dates: First submitted 2015-07-20; First posted 2015-10-05 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK2269557; Asthma; Pharmacokinetics; Safety; Adults; DISKUS Dry Powder Inhaler; Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2269557 and Placebo (Experimental): Each subject will complete two treatment periods: GSK2269557 1000 mcg in one treatment period, and matching placebo in the other treatment period. Each treatment will be administered once daily for 28 days (+/- 2 days) via the DISKUS DPI. The treatment periods will be separated by a washout of at least 4 weeks.
  Interventions: Drug: GSK2269557 DPI; Drug: Placebo DPI

INTERVENTIONS:
Drug: GSK2269557 DPI — GSK2269557 will be supplied as a lactose blend in a DISKUS DPI with a unit dose strength of 500 mcg. 2 inhalations will be taken every morning before breakfast.
Drug: Placebo DPI — Placebo will be lactose in a DISKUS DPI. 2 inhalations will be taken every morning before breakfast.

SUMMARY:
This study is a multi-centre, randomised, double-blind, placebo-controlled (with rescue medication), two period crossover study in subjects with persistent uncontrolled asthma, currently not treated with an inhaled corticosteroid (ICS) or long acting beta 2 agonist (LABA). This study is the first administration of GSK2269557 to asthmatic subjects, and the aims of the study are to investigate the efficacy, safety, tolerability, and pharmacokinetics of four weeks of treatment with orally inhaled GSK2269557 1000 microgram (mcg) in subjects with persistent uncontrolled asthma. In a sub-study, biological mediators will be measured from induced sputum and blood.

Approximately 50 subjects will be randomised into the study (including approximately 16 subjects in the sputum sub-study). Each subject will complete two treatment periods: subjects will be randomised to receive GSK2269557 1000 mcg in one treatment period, and matching placebo in the other treatment period. Each treatment will be administered once daily for 28 days (+/- 2 days) via the DISKUS™ dry powder inhaler (DPI).

The study will consist of a Screening Visit; a Run-in Period (approximately 2 weeks in duration); two 28-day Treatment Periods (each with 4 clinic visits); a 4-week Washout Period (between the Treatment Periods); and a Follow-up Visit. The total duration of the study for each subject will be approximately 16 weeks. DISKUS is a registered trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with an intermittent short acting beta 2 agonist (SABA) or other non-corticosteroid controllers. Non corticosteroid controllers (e.g. leukotriene receptor antagonists [LTRAs]) must be discontinued from Screening until the end of Treatment Period 2.
* Able to replace current SABA treatment with salbutamol metered dose inhaler (MDI) at Screening for use as needed for the duration of the study. Judged capable of withholding salbutamol for at least 4 hours prior to FEV1 assessments.
* No use of an ICS or LABA for at least 12 weeks prior to first dose of study medication.
* A best pre-bronchodilator FEV1 >=60 percent (%) of the predicted normal value at screening.
* FEV1 increase by >=12% and >=200 milliliter (mL) over baseline value within 10-40 minutes of inhalation of 400 mcg salbutamol MDI (a spacer device may be used if required).
* Positive skin prick test to common aero-allergen(s) at screening (not historical).
* Sputum sub-study only: Able to produce >100 milligram (mg) of sputum at screening or during the run-in period.
* Body weight >=45 kilogram (kg) and body mass index (BMI) within the range 18-32 kilogram per meter square (kg/m^2) (inclusive).
* Male subject: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the first dose of study medication until completion of the follow-up visit.

  1. Vasectomy with documentation of azoospermia.
  2. Male condom plus partner use of one of the contraceptive options below:

Contraceptive subdermal implant with a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system with a <1% rate of failure per year, as stated in the product label; Oral contraceptive, either combined or progestogen alone, injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches.

* Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

  1. Non-reproductive potential defined as pre-menopausal females with one of the following: Documented tubal ligation Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion Hysterectomy Documented bilateral oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  2. Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) modified list of highly effective methods for avoiding pregnancy in females of reproductive potential (FRP) requirements from 30 days prior to the first dose of study medication and until completion of the follow-up visit.

Contraceptive subdermal implant that meets the effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral contraceptive, either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject; Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository).

This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the consent form and the protocol. The informed consent must be signed prior to any study related procedure, including change in asthma medication.

Exclusion Criteria:

* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* Any severe asthma exacerbation, defined as deterioration of asthma requiring the use of systemic corticosteroids (oral, parenteral or depot) within 12 weeks of screening, or an inpatient hospitalisation or emergency department visit due to asthma that required systemic corticosteroids within 6 months of screening.
* Respiratory Infection: culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that has not resolved within 4 weeks of screening and led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Concurrent Respiratory Disease: current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, lung cancer, or other respiratory abnormalities other than asthma.
* Alanine aminotransferase (ALT) >2x upper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc >450 millisecond (msec) or QTc >480 msec in subjects with bundle branch block.
* Other laboratory abnormalities or concurrent diseases/clinical: clinically significant laboratory abnormality, uncontrolled condition or disease state that, in the opinion of the investigator (in consultation with the GSK Medical Monitor, if required), would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
* Use of any of the prohibited medications listed in the protocol.
* Current smokers or subjects with a history of smoking within 6 months of screening, or with a total pack year history of >5 pack years.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof (including lactose) or a history of drug or other allergy (including a milk protein allergy) that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Sputum sub-study only: History of sensitivity to the induced sputum procedure.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dose of study medication in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dose of study medication.
* Affiliation with investigator site: subject is an investigator; sub-investigator; study co-ordinator; employee of a participating investigator or study site; or, an immediate family member of the aforementioned, that is involved in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-01; Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Germany (8):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Magdeburg

REFERENCES:
- [Derived] Khindri S, Cahn A, Begg M, Montembault M, Leemereise C, Cui Y, Hogg A, Wajdner H, Yang S, Robertson J, Hamblin JN, Ludwig-Sengpiel A, Kornmann O, Hessel EM. A Multicentre, Randomized, Double-Blind, Placebo-Controlled, Crossover Study To Investigate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Repeat Doses of Inhaled Nemiralisib in Adults with Persistent, Uncontrolled Asthma. J Pharmacol Exp Ther. 2018 Dec;367(3):405-413. doi: 10.1124/jpet.118.249516. Epub 2018 Sep 14. PMID 30217958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants entered the 2 week Run-in phase and participants who met the randomization eligibility criteria entered into the 4 week Double-blind treatment period (DBTP) 1 followed by a 4-week wash-out period, 4 weeks DBTP 2 and a 2 week follow-up phase. The total duration of participation in the study was 16 weeks.
Pre-assignment Details: A total of 108 participants with persistent uncontrolled asthma, currently not treated with an inhaled corticosteroid (ICS) or long acting beta2 agonist (LABA) were screened, of these, 58 were screen failures and 50 entered the Run-in phase. All 50 par. were randomized into the study and received study treatments.
Groups:
- Placebo, Then GSK2269557: Participants received placebo drug once daily via dry powder inhaler for 28 days during Treatment Period 1. After a washout period of 4 weeks, participants received GSK2269557 1000 micrograms (µg) drug once daily via dry powder inhaler for 28 days during Treatment Period 2. In addition, salbutamol was provided to participants to use on an as-needed basis for relief of asthma symptoms.
- GSK2269557, Then Placebo: Participants received GSK2269557 1000 µg drug once daily via dry powder inhaler for the 28 days during Treatment Period 1. After a washout period of 4 weeks, participants received placebo drug once daily via dry powder inhaler for 28 days during Treatment Period 2. In addition, salbutamol was provided to participants to use on an as-needed basis for relief of asthma symptoms.
Period: Treatment Period 1 (Up to 4 Weeks)
Arm/Group | Placebo, Then GSK2269557 | GSK2269557, Then Placebo
Started | 24 | 26
Completed | 22 | 23
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Other: Reached stopping criteria | 2 | 0
Period: Washout Period (Up to 4 Weeks)
Arm/Group | Placebo, Then GSK2269557 | GSK2269557, Then Placebo
Started | 22 | 23
Completed | 22 | 23
Not Completed | 0 | 0
Period: Treatment Period 2 (Up to 4 Weeks)
Arm/Group | Placebo, Then GSK2269557 | GSK2269557, Then Placebo
Started | 22 | 23
Completed | 22 | 20
Not Completed | 0 | 3
Not completed — Other: Reached stopping criteria | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: In Sequence 1 participants received placebo drug once daily via dry powder inhaler for 28 days during Treatment Period 1. After a washout period of 4 weeks, participants received GSK2269557 1000 micrograms (µg) drug once daily via dry powder inhaler for 28 days during Treatment Period 2. In addition, salbutamol was provided to participants to use on an as-needed basis for relief of asthma symptoms. In Sequence 2 participants received GSK2269557 1000 micrograms (µg) drug once daily via dry powder inhaler for 28 days during Treatment Period 1. After a washout period of 4 weeks, participants received placebo drug once daily via dry powder inhaler for 28 days during Treatment Period 2. In addition, salbutamol was provided to participants to use on an as-needed basis for relief of asthma symptoms.
Arm/Group | All Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European Heritage | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Day 28 in Intent-To-Treat (ITT) Population
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is the maximum volume of air that can be forced out in one second after taking a deep breath approximately 24 hours after the last administration of study drug. FEV1 was measured using a spirometer. Change from Baseline is calculated as post-Baseline value minus Baseline value where Baseline is defined as Day 1 (pre-dose).
Time Frame: Baseline and Day 28 for each treatment period
Population: The analysis was performed on the ITT Population which comprised of all participants who received at least one dose of trial medication and have at least one post-dose efficacy assessment. Six participants had entered the study without spirometric evidence of disease, and were excluded from the ITT population prior to unblinding.
Measure: Median (95% Confidence Interval); unit: Liters
Groups:
- Placebo: Participants who received matching placebo once daily via dry powder inhaler for 28 days in either treatment period 1 or 2.
- GSK2269557 1000 µg: Participants who received GSK2269557 1000 µg once daily via dry powder inhaler for 28 days in either treatment period 1 or 2.
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 37 | 39
Liters | 0.027 [-0.066 to 0.117] | 0.035 [-0.061 to 0.124]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.57, Bayesian repeated measures model. — The data entered for the p-value represents the posterior probability that the true treatment difference is greater than zero; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference. = 0.007, 95% CI 2-sided [-0.083 to 0.102], Standard Deviation 0.0468 — The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median difference is calculated as GSK2269557 1000 μg minus Placebo

2. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Day 28 in Per Protocol (PP) Population
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is the maximum volume of air that can be forced out in one second after taking a deep breath approximately 24 hours after the last administration of study drug. FEV1 was measured using a spirometer. Change from Baseline is calculated as post-Baseline value minus Baseline value where Baseline is defined as Day 1 (pre-dose). The analysis was performed on the PP Population which comprised of all participants in the ITT Population not identified as major protocol violators.
Time Frame: Baseline and Day 28 for each treatment period
Population: PP Population
Measure: Median (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 35 | 37
Liters | 0.029 [-0.073 to 0.119] | 0.042 [-0.058 to 0.132]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.61, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference. = 0.013, 95% CI 2-sided [-0.084 to 0.113], Standard Deviation 0.0501 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Weighted Mean (0-4 Hours) FEV1 at Day 28
Description: The weighted mean FEV1 on Day 28 was calculated using data collected pre-dose and at 1 hour, 2 hours, 3 hours, and 4 hours post-dose. The weighted mean FEV1 was derived by calculating the average area under the curve using the trapezoidal rule, and then dividing by the relevant time interval.
Time Frame: Day 28 for each treatment period
Population: ITT Population. Only those participants with data available at specific time point were analyzed.
Measure: Median (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 38 | 40
Liters | 2.672 [2.556 to 2.783] | 2.722 [2.607 to 2.836]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other — The data entered for the p-value represents the posterior probability that the true treatment difference is greater than zero; p = 0.731, Bayesian model; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.050, 95% CI 2-sided [-0.111 to 0.210], Standard Deviation 0.0818 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Trough FEV1 at Day 7 and Day 14
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The trough FEV1 is the maximum volume of air that can be forced out in one second after taking a deep breath approximately 24 hrs after the last administration of study drug. Change from Baseline values were calculated as post-Baseline values minus Baseline value where Baseline was defined as Day 1 (pre-dose). The number of participants with data available at the specified time points are represented by n=X in the category titles.
Time Frame: Baseline, Day 7 and Day 14 for each treatment period
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Liters
  Day 7; n= 39, 40: number analyzed (Participants) | 39 | 40
  Day 7; n= 39, 40 | 0.012 [-0.102 to 0.131] | 0.003 [-0.113 to 0.119]
  Day 14; n= 38,41: number analyzed (Participants) | 38 | 41
  Day 14; n= 38,41 | 0.016 [-0.086 to 0.116] | 0.040 [-0.061 to 0.137]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.44, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = -0.009, 95% CI 2-sided [-0.151 to 0.131], Standard Deviation 0.0712 — Day 7. The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median difference is calculated as GSK2269557 1000 μg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.66, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.024, 95% CI 2-sided [-0.087 to 0.137], Standard Deviation 0.0570 — Day 14. The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median difference is calculated as GSK2269557 1000 μg minus Placebo

5. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Day 7, Day 14 and Day 28
Description: FVC is defined as the total amount of air exhaled during the FEV test. Data was collected pre-dose at Baseline (Day 1), Day 7, Day 14 and Day 28. Change from Baseline was calculated as the post-Baseline value minus the Baseline value where Baseline was defined as Day 1 (pre-dose). The number of participants with data available at the specified time points are represented by n=X in the category titles.
Time Frame: Baseline, Day 7, Day 14 and Day 28 for each treatment period
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Liter
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Liter
  Day 7; n= 39,40: number analyzed (Participants) | 39 | 40
  Day 7; n= 39,40 | 0.036 [-0.075 to 0.146] | 0.015 [-0.097 to 0.126]
  Day 14; n= 38,41: number analyzed (Participants) | 38 | 41
  Day 14; n= 38,41 | -0.002 [-0.110 to 0.107] | 0.038 [-0.069 to 0.146]
  Day 28; n= 37,39: number analyzed (Participants) | 37 | 39
  Day 28; n= 37,39 | 0.017 [-0.092 to 0.124] | 0.054 [-0.052 to 0.159]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.35, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = -0.021, 95% CI 2-sided [-0.140 to 0.099], Standard Deviation 0.0609 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.76, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.040, 95% CI 2-sided [-0.071 to 0.156], Standard Deviation 0.0578 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.76, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.038, 95% CI 2-sided [-0.073 to 0.148], Standard Deviation 0.0559 — Day 28. The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median difference is calculated as GSK2269557 1000 μg minus Placebo

6. Secondary Outcome: Change From Baseline in FEV1/FVC at Day 7, Day 14 and Day 28
Description: FEV1 and FVC are measures of lung function. FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the total amount of air exhaled during the FEV test. Change from Baseline in FEV1/FVC at Day 7, Day 14 and Day 28 was calculated as post-Baseline value minus Baseline value where Baseline was defined as Day 1 (pre-dose). The number of participants with data available at the specified time points are represented by n=X in the category titles.
Time Frame: Baseline, Day 7, Day 14 and Day 28 for each treatment period
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Percentage of exhaled air
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Percentage of exhaled air
  Day 7; n= 39,40: number analyzed (Participants) | 39 | 40
  Day 7; n= 39,40 | -0.956 [-2.337 to 0.495] | -0.855 [-2.285 to 0.517]
  Day 14; n= 38,41: number analyzed (Participants) | 38 | 41
  Day 14; n= 38,41 | -0.456 [-1.944 to 0.986] | -0.444 [-1.899 to 0.992]
  Day 28; n= 37,39: number analyzed (Participants) | 37 | 39
  Day 28; n= 37,39 | -0.691 [-2.050 to 0.638] | -0.791 [-2.163 to 0.516]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.56, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.083, 95% CI 2-sided [-1.102 to 1.346], Standard Deviation 0.6175 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.51, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.014, 95% CI 2-sided [-1.271 to 1.341], Standard Deviation 0.6672 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.41, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = -0.113, 95% CI 2-sided [-1.125 to 0.908], Standard Deviation 0.5148 — [estimate comment as in outcome 5, analysis 3]

7. Secondary Outcome: Change From Baseline in Asthma Control Test (ACT) Score at Day 28
Description: The total ACT score is the sum of five-item questionnaires developed as a measurement of asthma control. Total score can range from five (worse control) to 25 (full control), with higher scores reflecting greater asthma control. Total ACT score at Day 1 (Baseline) and Day 28 in both Treatment Periods was used for this analysis. Change from Baseline in ACT was calculated as post-Baseline value minus Baseline value where Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline and Day 28 for each treatment period
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 38 | 40
Score on a scale | 1.4 [0.5 to 2.2] | 1.9 [1.0 to 2.7]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.81, Bayesian model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median difference = 0.5, 95% CI 2-sided [-0.6 to 1.7], Standard Deviation 0.59 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Daily FEV1 Averaged Over the Treatment Period
Description: Triplicate measurements of FEV1 were collected in an eDiary pre-dose before breakfast [ante meridiem (AM)], and approximately 12 hours later at evening [post-meridiem (PM)]. The average change from Baseline was calculated by summing the total value of the endpoint (i.e. change from Baseline) within the time period of interest and dividing by the number of days with non-missing data for that endpoint to obtain an average for each subject. The AM Baseline is the Day 1 AM value, the PM Baseline is the last PM reading prior to taking the first dose of blinded study medication within that Treatment Period. The number of participants with data available at the specified time points are represented by n=X in the category titles.
Time Frame: Baseline and up to Day 28 for each treatment period
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Liter
  AM; n= 38, 40: number analyzed (Participants) | 38 | 40
  AM; n= 38, 40 | 0.000 (0.2019) | 0.065 (0.2974)
  PM; n= 34, 39: number analyzed (Participants) | 34 | 39
  PM; n= 34, 39 | 0.013 (0.2634) | 0.115 (0.3802)

9. Secondary Outcome: Change From Baseline in Daily Peak Expiratory Flow (PEF) Averaged Over the Treatment Period
Description: Triplicate measurements of PEF were collected in an eDiary pre-dose before breakfast (AM), and approximately 12 hours later at evening (PM). The average change from Baseline was calculated by summing the total value of the endpoint (i.e. change from Baseline) within the time period of interest and dividing by the number of days with non-missing data for that endpoint to obtain an average for each subject. The AM Baseline is the Day 1 AM value, the PM Baseline is the last PM reading prior to taking the first dose of blinded study medication within that Treatment Period. The number of participants with data available at the specified time points are represented by n=X in the category titles.
Time Frame: Baseline and up to Day 28 for each treatment period
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Liter/minute
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Liter/minute
  AM; n= 38,40: number analyzed (Participants) | 38 | 40
  AM; n= 38,40 | -4.8 (32.44) | 14.2 (46.11)
  PM; n= 34, 39: number analyzed (Participants) | 34 | 39
  PM; n= 34, 39 | 9.8 (36.05) | 29.8 (64.28)

10. Secondary Outcome: Change From Baseline in Trough Fractional Exhaled Nitric Oxide (FeNO) at Day 7, Day 14 and Day 28
Description: Participants with asthma have high levels of NO in their exhaled breath. Evaluation of FeNO is a quantitative, noninvasive method of measuring airway inflammation to assess airway diseases including asthma. FeNO was measured in the clinic using a handheld electronic device. Change from Baseline for Day 7, Day 14 and Day 28 was calculated as the post-Baseline value minus the Baseline value where Baseline was defined as Day 1 (pre-dose). The number of participants with data available at the specified time points are represented by n=X in the category titles.
Time Frame: Baseline, Day 7, Day 14 and Day 28 for each treatment period
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Part per billion (PPB)
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Part per billion (PPB)
  Day 7; n= 38,34: number analyzed (Participants) | 38 | 34
  Day 7; n= 38,34 | 1.03 [0.93 to 1.13] | 0.91 [0.82 to 1.01]
  Day 14; n= 34,35: number analyzed (Participants) | 34 | 35
  Day 14; n= 34,35 | 0.99 [0.89 to 1.11] | 0.95 [0.85 to 1.05]
  Day 28; n= 34,34: number analyzed (Participants) | 34 | 34
  Day 28; n= 34,34 | 1.03 [0.91 to 1.17] | 1.03 [0.91 to 1.17]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.97, Bayesian repeated measures model — The data entered for the p-value represents the posterior probability that the true treatment ratio is less than 1; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median ratio = 0.89, 95% CI 2-sided [0.78 to 1.00], Standard Deviation 0.063 — Day 7. The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median ratio is calculated as GSK2269557 1000 μg/ Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.76, Bayesian repeated measures model — The data entered for the p-value represents the posterior probability that the true treatment ratio is less than 1; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median ratio = 0.95, 95% CI 2-sided [0.83 to 1.09], Standard Deviation 0.071 — Day 14. The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median ratio is calculated as GSK2269557 1000 μg/ Placebo
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Other; p = 0.51, Bayesian repeated measures model — The data entered for the p-value represents the posterior probability that the true treatment ratio is less than one; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted; Posterior median ratio = 1.00, 95% CI 2-sided [0.84 to 1.18], Standard Deviation 0.085 — Day 28. The data entered as the 95% confidence interval represents the 95% equi-tailed credible interval. The posterior median ratio is calculated as GSK2269557 1000 μg/ Placebo

11. Secondary Outcome: Mean Number of Inhalations Per Day of Rescue Medication (Salbutamol) Over the Treatment Period
Description: Daily recordings of rescue medication use were collected in an eDiary by participants. The mean number of inhalations per day of rescue medication was calculated for each participant as number of inhalations over the time period of interest divided by number of days when rescue medication was taken over the time period of interest.
Time Frame: Up to Day 28 for each treatment period
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Inhalations/day
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 38 | 39
Inhalations/day | 3.0 (1.86) | 2.7 (1.53)

12. Secondary Outcome: Percentage of Rescue Free Days Over the Treatment Period
Description: Daily recordings of rescue medication use were collected in an eDiary by participants. Percentage of rescue free days was calculated as the number of rescue free days divided by length of treatment period.
Time Frame: Up to Day 28 for each treatment period
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 42 | 42
Percentage of days | 49.5 (35.04) | 47.3 (34.79)

13. Secondary Outcome: Number of Participants With On-treatment Serious Adverse Events (SAEs) and Non-serious Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The analysis was performed on Safety Population which comprised of all participants who were randomized into the study.
Time Frame: From the Start of IP up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 47 | 48
Participants
  non-SAE | 13 | 19
  SAE | 0 | 0

14. Secondary Outcome: Number of Participants With Abnormal Values of Clinical Chemistry Parameters
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters by Potential Clinical Importance Criteria. The clinical chemistry parameters included albumin, calcium, creatinine, glucose, potassium and sodium. Participants were counted in the category that their value changes to (low, normal or high), unless there is no change in their category. The number of participants with data available at the specified data points are represented by n=X in the category titles.
Time Frame: From start of IP up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 47 | 48
Participants
  Albumin; Day 1; Change to low; n= 47, 48 | 0 | 0
  Albumin; Day 14; Change to low; n= 42, 48: number analyzed (Participants) | 42 | 48
  Albumin; Day 14; Change to low; n= 42, 48 | 0 | 0
  Albumin; Day 28; Change to low; n= 41, 45: number analyzed (Participants) | 41 | 45
  Albumin; Day 28; Change to low; n= 41, 45 | 0 | 0
  Calcium; Day 1; Change to low; n= 47, 48 | 0 | 0
  Calcium; Day 1; Change to high; n= 47, 48 | 0 | 0
  Calcium; Day 14; Change to low; n= 42, 48: number analyzed (Participants) | 42 | 48
  Calcium; Day 14; Change to low; n= 42, 48 | 0 | 0
  Calcium; Day 14; Change to high; n= 42, 48: number analyzed (Participants) | 42 | 48
  Calcium; Day 14; Change to high; n= 42, 48 | 0 | 0
  Calcium; Day 28; Change to high; n= 40, 45: number analyzed (Participants) | 40 | 45
  Calcium; Day 28; Change to high; n= 40, 45 | 0 | 0
  Calcium; Day 28; Change to low; n= 40, 45: number analyzed (Participants) | 40 | 45
  Calcium; Day 28; Change to low; n= 40, 45 | 0 | 0
  Glucose; Day 1; Change to low; n= 47, 48 | 0 | 0
  Glucose; Day 1; change to high; n= 47, 48 | 0 | 0
  Glucose; Day 14; Change to low; n= 42, 48: number analyzed (Participants) | 42 | 48
  Glucose; Day 14; Change to low; n= 42, 48 | 1 | 0
  Glucose; Day 14; change to high; n= 42, 48: number analyzed (Participants) | 42 | 48
  Glucose; Day 14; change to high; n= 42, 48 | 0 | 0
  Glucose; Day 28; Change to low; n= 41, 45: number analyzed (Participants) | 41 | 45
  Glucose; Day 28; Change to low; n= 41, 45 | 0 | 0
  Glucose; Day 28; Change to high; n= 41, 45: number analyzed (Participants) | 41 | 45
  Glucose; Day 28; Change to high; n= 41, 45 | 0 | 0
  Potassium; Day 1; Change to low; n= 47, 48 | 0 | 0
  Potassium; Day 1; Change to high; n= 47, 48 | 0 | 0
  Potassium; Day 14; Change to low; n= 42, 48: number analyzed (Participants) | 42 | 48
  Potassium; Day 14; Change to low; n= 42, 48 | 0 | 0
  Potassium; Day 14; Change to high; n= 42, 48: number analyzed (Participants) | 42 | 48
  Potassium; Day 14; Change to high; n= 42, 48 | 0 | 0
  Potassium; Day 28; Change to low; n= 40, 45: number analyzed (Participants) | 40 | 45
  Potassium; Day 28; Change to low; n= 40, 45 | 0 | 0
  Potassium; Day 28; Change to high; n= 40, 45: number analyzed (Participants) | 40 | 45
  Potassium; Day 28; Change to high; n= 40, 45 | 0 | 0
  Sodium; Day 1; Change to low; n= 47, 48 | 0 | 0
  Sodium; Day 1; Change to high; n= 47, 48 | 0 | 0
  Sodium; Day 14; Change to low; n= 42, 48: number analyzed (Participants) | 42 | 48
  Sodium; Day 14; Change to low; n= 42, 48 | 0 | 0
  Sodium; Day 14; Change to high; n= 42, 48: number analyzed (Participants) | 42 | 48
  Sodium; Day 14; Change to high; n= 42, 48 | 0 | 0
  Sodium; Day 28; Change to low; n= 41, 45: number analyzed (Participants) | 41 | 45
  Sodium; Day 28; Change to low; n= 41, 45 | 0 | 0
  Sodium; Day 28; Change to high; n= 41, 45: number analyzed (Participants) | 41 | 45
  Sodium; Day 28; Change to high; n= 41, 45 | 0 | 0
  Hematocrit; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  Hematocrit; Day 1; Change to high; n= 46, 47 | 0 | 0
  Hematocrit; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  Hematocrit; Day 14; Change to high; n= 43, 47 | 0 | 0
  Hematocrit; Day 28; Change to high; n= 42, 44: number analyzed (Participants) | 42 | 44
  Hematocrit; Day 28; Change to high; n= 42, 44 | 0 | 0
  Hemoglobin; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  Hemoglobin; Day 1; Change to high; n= 46, 47 | 0 | 0
  Hemoglobin; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  Hemoglobin; Day 14; Change to high; n= 43, 47 | 0 | 0
  Hemoglobin; Day 28; Change to high; n= 42, 44: number analyzed (Participants) | 42 | 44
  Hemoglobin; Day 28; Change to high; n= 42, 44 | 0 | 0
  Lymphocytes; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  Lymphocytes; Day 1; Change to low; n= 46, 47 | 0 | 0
  Lymphocytes; Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  Lymphocytes; Day 14; Change to low; n= 43, 47 | 0 | 0
  Lymphocytes; Day 28; Change to low; n= 42, 44: number analyzed (Participants) | 42 | 44
  Lymphocytes; Day 28; Change to low; n= 42, 44 | 0 | 0
  Platelet count; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  Platelet count; Day 1; Change to low; n= 46, 47 | 0 | 0
  Platelet count; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  Platelet count; Day 1; Change to high; n= 46, 47 | 0 | 0
  Platelet count; Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  Platelet count; Day 14; Change to low; n= 43, 47 | 0 | 0
  Platelet count; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  Platelet count; Day 14; Change to high; n= 43, 47 | 0 | 0
  Platelet count; Day 28; Change to low; n= 42, 43: number analyzed (Participants) | 42 | 43
  Platelet count; Day 28; Change to low; n= 42, 43 | 0 | 0
  Platelet count; Day 28; Change to high; n= 42, 43: number analyzed (Participants) | 42 | 43
  Platelet count; Day 28; Change to high; n= 42, 43 | 0 | 0
  Total neutrophils; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  Total neutrophils; Day 1; Change to low; n= 46, 47 | 0 | 0
  Total neutrophils;Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  Total neutrophils;Day 14; Change to low; n= 43, 47 | 0 | 1
  Total neutrophils; Day 28; Change to low; n= 42,44: number analyzed (Participants) | 42 | 44
  Total neutrophils; Day 28; Change to low; n= 42,44 | 0 | 0
  WBC; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  WBC; Day 1; Change to low; n= 46, 47 | 0 | 0
  WBC; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  WBC; Day 1; Change to high; n= 46, 47 | 0 | 0
  WBC; Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  WBC; Day 14; Change to low; n= 43, 47 | 0 | 0
  WBC; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  WBC; Day 14; Change to high; n= 43, 47 | 0 | 0
  WBC; Day 28; Change to low; n= 42, 44: number analyzed (Participants) | 42 | 44
  WBC; Day 28; Change to low; n= 42, 44 | 0 | 0
  WBC; Day 28; Change to high; n= 42, 44: number analyzed (Participants) | 42 | 44
  WBC; Day 28; Change to high; n= 42, 44 | 0 | 0

15. Secondary Outcome: Number of Participants With Abnormal Values of Hematology Parameters
Description: Blood samples were collected from participants for evaluation of hematology parameters by Potential Clinical Importance Criteria. The hematology parameters included hematocrit, hemoglobin, lymphocytes, total neutrophils, platelets and white blood cells (WBC). Participants were counted in the category that their value changes to (low, normal or high), unless there is no change in their category. The number of participants with data available at the specified data points are represented by n=X in the category titles.
Time Frame: From start of IP up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 47 | 48
Participants
  Hematocrit; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  Hematocrit; Day 1; Change to high; n= 46, 47 | 0 | 0
  Hematocrit; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  Hematocrit; Day 14; Change to high; n= 43, 47 | 0 | 0
  Hematocrit; Day 28; Change to high; n= 42, 44: number analyzed (Participants) | 42 | 44
  Hematocrit; Day 28; Change to high; n= 42, 44 | 0 | 0
  Hemoglobin; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  Hemoglobin; Day 1; Change to high; n= 46, 47 | 0 | 0
  Hemoglobin; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  Hemoglobin; Day 14; Change to high; n= 43, 47 | 0 | 0
  Hemoglobin; Day 28; Change to high; n= 42, 44: number analyzed (Participants) | 42 | 44
  Hemoglobin; Day 28; Change to high; n= 42, 44 | 0 | 0
  Lymphocytes; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  Lymphocytes; Day 1; Change to low; n= 46, 47 | 0 | 0
  Lymphocytes; Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  Lymphocytes; Day 14; Change to low; n= 43, 47 | 0 | 0
  Lymphocytes; Day 28; Change to low; n= 42, 44: number analyzed (Participants) | 42 | 44
  Lymphocytes; Day 28; Change to low; n= 42, 44 | 0 | 0
  Platelet count; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  Platelet count; Day 1; Change to low; n= 46, 47 | 0 | 0
  Platelet count; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  Platelet count; Day 1; Change to high; n= 46, 47 | 0 | 0
  Platelet count; Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  Platelet count; Day 14; Change to low; n= 43, 47 | 0 | 0
  Platelet count; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  Platelet count; Day 14; Change to high; n= 43, 47 | 0 | 0
  Platelet count; Day 28; Change to low; n= 42, 43: number analyzed (Participants) | 42 | 43
  Platelet count; Day 28; Change to low; n= 42, 43 | 0 | 0
  Platelet count; Day 28; Change to high; n= 42, 43: number analyzed (Participants) | 42 | 43
  Platelet count; Day 28; Change to high; n= 42, 43 | 0 | 0
  Total neutrophils; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  Total neutrophils; Day 1; Change to low; n= 46, 47 | 0 | 0
  Total neutrophils;Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  Total neutrophils;Day 14; Change to low; n= 43, 47 | 0 | 1
  Total neutrophils; Day 28; Change to low; n= 42,44: number analyzed (Participants) | 42 | 44
  Total neutrophils; Day 28; Change to low; n= 42,44 | 0 | 0
  WBC; Day 1; Change to low; n= 46, 47: number analyzed (Participants) | 46 | 47
  WBC; Day 1; Change to low; n= 46, 47 | 0 | 0
  WBC; Day 1; Change to high; n= 46, 47: number analyzed (Participants) | 46 | 47
  WBC; Day 1; Change to high; n= 46, 47 | 0 | 0
  WBC; Day 14; Change to low; n= 43, 47: number analyzed (Participants) | 43 | 47
  WBC; Day 14; Change to low; n= 43, 47 | 0 | 0
  WBC; Day 14; Change to high; n= 43, 47: number analyzed (Participants) | 43 | 47
  WBC; Day 14; Change to high; n= 43, 47 | 0 | 0
  WBC; Day 28; Change to low; n= 42, 44: number analyzed (Participants) | 42 | 44
  WBC; Day 28; Change to low; n= 42, 44 | 0 | 0
  WBC; Day 28; Change to high; n= 42, 44: number analyzed (Participants) | 42 | 44
  WBC; Day 28; Change to high; n= 42, 44 | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormal Vital Sign Values
Description: Number of participants with abnormal values of vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate were evaluated. Vital signs outside the range of potential clinical importance are presented at the indicated timepoints: Day 7, Day 14, Day 28 and follow-up/Early withdrawal. The number of participants with data available at the specified data points are represented by n=X in the category titles.
Time Frame: From start of IP up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 47 | 48
Participants
  DBP; Day 7; Change to low; n= 46, 46: number analyzed (Participants) | 46 | 46
  DBP; Day 7; Change to low; n= 46, 46 | 0 | 0
  DBP; Day 7; Change to high; n= 46, 46: number analyzed (Participants) | 46 | 46
  DBP; Day 7; Change to high; n= 46, 46 | 0 | 0
  DBP; Day 14; Change to low; n= 43, 48: number analyzed (Participants) | 43 | 48
  DBP; Day 14; Change to low; n= 43, 48 | 0 | 0
  DBP; Day 14; Change to high; n= 43, 48: number analyzed (Participants) | 43 | 48
  DBP; Day 14; Change to high; n= 43, 48 | 1 | 0
  DBP; Day 28; Change to low; n= 42, 45: number analyzed (Participants) | 42 | 45
  DBP; Day 28; Change to low; n= 42, 45 | 0 | 0
  DBP; Day 28; Change to high; n= 42, 45: number analyzed (Participants) | 42 | 45
  DBP; Day 28; Change to high; n= 42, 45 | 0 | 1
  SBP; Day 7; Change to low; n= 46, 46: number analyzed (Participants) | 46 | 46
  SBP; Day 7; Change to low; n= 46, 46 | 0 | 0
  SBP; Day 7; Change to high; n= 46, 46: number analyzed (Participants) | 46 | 46
  SBP; Day 7; Change to high; n= 46, 46 | 0 | 0
  SBP; Day 14; Change to low; n= 43, 48: number analyzed (Participants) | 43 | 48
  SBP; Day 14; Change to low; n= 43, 48 | 0 | 0
  SBP; Day 14; Change to high; n= 43, 48: number analyzed (Participants) | 43 | 48
  SBP; Day 14; Change to high; n= 43, 48 | 1 | 0
  SBP; Day 28; Change to low; n= 42, 45: number analyzed (Participants) | 42 | 45
  SBP; Day 28; Change to low; n= 42, 45 | 0 | 0
  SBP; Day 28; Change to high; n= 42, 45: number analyzed (Participants) | 42 | 45
  SBP; Day 28; Change to high; n= 42, 45 | 0 | 0
  Heart rate; Day 7; Change to low; n= 46, 46: number analyzed (Participants) | 46 | 46
  Heart rate; Day 7; Change to low; n= 46, 46 | 0 | 0
  Heart rate; Day 7; Change to high; n= 46, 46: number analyzed (Participants) | 46 | 46
  Heart rate; Day 7; Change to high; n= 46, 46 | 0 | 0
  Heart rate; Day 14; Change to low; n= 43, 48: number analyzed (Participants) | 43 | 48
  Heart rate; Day 14; Change to low; n= 43, 48 | 0 | 0
  Heart rate; Day 14; Change to high; n= 43, 48: number analyzed (Participants) | 43 | 48
  Heart rate; Day 14; Change to high; n= 43, 48 | 0 | 0
  Heart rate; Day 28; Change to low; n= 42, 45: number analyzed (Participants) | 42 | 45
  Heart rate; Day 28; Change to low; n= 42, 45 | 0 | 0
  Heart rate; Day 28; Change to high; n= 42, 45: number analyzed (Participants) | 42 | 45
  Heart rate; Day 28; Change to high; n= 42, 45 | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single measurements of 12-lead ECGs were obtained after 5 minutes rest in a semi-supine position at Baseline (Day 1 pre dose) , Day 7, Day 28 pre-dose in each treatment period using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc). ECG values were recorded as abnormal not clinically significant (NCS) and abnormal clinically significant (CS). The number of participants with data available at the specified data points are represented by n= X in the category titles.
Time Frame: Up to Day 28 for each treatment period
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 47 | 48
Participants
  Day 1; abnormal NCS; n= 47,48 | 2 | 5
  Day 1; abnormal CS; n= 47,48 | 0 | 0
  Day 7; abnormal NCS; n= 46,46: number analyzed (Participants) | 46 | 46
  Day 7; abnormal NCS; n= 46,46 | 1 | 4
  Day 7; abnormal CS; n= 46,46: number analyzed (Participants) | 46 | 46
  Day 7; abnormal CS; n= 46,46 | 0 | 0
  Day 28; abnormal NCS; n= 42, 45: number analyzed (Participants) | 42 | 45
  Day 28; abnormal NCS; n= 42, 45 | 0 | 3
  Day 28; abnormal CS; n= 42,45: number analyzed (Participants) | 42 | 45
  Day 28; abnormal CS; n= 42,45 | 0 | 0
  Any time Post-Baseline; abnormal NCS; n= 47,48 | 1 | 6
  Any time Post Baseline; abnormal CS; n= 47,48 | 0 | 0

18. Secondary Outcome: Plasma Concentration of GSK2269557
Description: Blood samples were collected from participants for pharmacokinetic (PK) analysis at Day 7, Day 14 and Day 28 pre dose. On Day 28 samples were also collected between 5-10 minutes post dose and between 2.5-3.5 hours post dose. The analysis was performed on PK Population which comprised of participants in the ITT Population for whom a PK sample was obtained and analyzed. The number of participants with data available at the specified data points are represented by n= X in the category titles.
Time Frame: Pre dose at Day 7 and Day 14. At Day 28 pre dose, 5-10 minutes and 2.5-3.5 hours post dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Picograms per Milliliter (Pg/mL)
Arm/Group | GSK2269557 1000 µg
Number analyzed (Participants) | 42
Picograms per Milliliter (Pg/mL)
  Day 7; pre dose; n= 40: number analyzed (Participants) | 40
  Day 7; pre dose; n= 40 | 555.7 [446.2 to 692.0]
  Day 14; pre dose; n= 40: number analyzed (Participants) | 40
  Day 14; pre dose; n= 40 | 520.7 [380.3 to 712.9]
  Day 28; pre dose; n= 38: number analyzed (Participants) | 38
  Day 28; pre dose; n= 38 | 649.2 [519.9 to 810.8]
  Day 28; 5-10 minutes post dose; n= 40: number analyzed (Participants) | 40
  Day 28; 5-10 minutes post dose; n= 40 | 1188.8 [990.5 to 1426.8]
  Day 28; 2.5-3.5 hours post dose; n= 40: number analyzed (Participants) | 40
  Day 28; 2.5-3.5 hours post dose; n= 40 | 1170.8 [976.1 to 1404.4]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment up to Week 14.
Description: Non-SAEs and SAEs were collected in Safety Population which comprised of all participants who were randomized.
Arm/Group | Placebo | GSK2269557 1000 µg
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 13/47 | 19/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | GSK2269557 1000 µg (N=48)
Nasopharyngitis (Infections and infestations) | 7 | 2
Headache (Nervous system disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.